CLINICAL TRIAL: NCT01410097
Title: Intentional Weight Reduction and Physical and Cognitive Function - A Look AHEAD Ancillary Study
Brief Title: Physical and Cognitive Function - Look AHEAD Ancillary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Pennington Biomedical Research Center (Other); University of Colorado, Denver (Other); University of Tennessee (Other); University of Pittsburgh (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00008777; R01AG033087 (NIH)
Record Dates: First submitted 2011-07-08; First posted 2011-08-04 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Weight Loss; Physical Function; Cognitive Function
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention (Experimental): Intensive Lifestyle Intervention that includes diet, physical activity, and behavior modification. The goal of the ILI intervention was for individuals to achieve and maintain a loss of at least 7% of initial body weight.
  Interventions: Behavioral: Lifestyle intervention
- Diabetes Support and Education (DSE) (Placebo Comparator): It offers an educational program to participants including developing support groups. Providing such benefits helps retain these participants in the trial.
  Interventions: Behavioral: Diabetes Support Education

INTERVENTIONS:
Behavioral: Lifestyle intervention — Intensive Lifestyle Intervention that includes diet, physical activity, and behavior modification. The goal of the ILI intervention was for individuals to achieve and maintain a loss of at least 7% of initial body weight.
  Arms: Lifestyle intervention
Behavioral: Diabetes Support Education — It offers an educational program to participants including developing support groups. Providing such benefits helps retain these participants in the trial.
  Arms: Diabetes Support and Education (DSE)

SUMMARY:
Obesity is associated with physical disability through both direct pathways (e.g., lower extremity pain, insufficient muscle strength) and indirect pathways (obesity-related comorbidities and inflammation). Furthermore, diabetes, a major obesity-related health condition, is associated with increased risk of disability and accelerated declines in physical and cognitive function. The investigators preliminary data suggest that intentional weight loss improves physical function, and there is strong circumstantial evidence that it would also benefit cognitive function.

To evaluate the role of intentional weight loss on physical and cognitive function, the investigators propose an ancillary study to the on-going Look AHEAD (Action for Health in Diabetes) trial. Look AHEAD is a multi-center, randomized clinical trial to examine the effects of a 4-year lifestyle intervention designed to achieve and maintain weight loss through decreased caloric intake and exercise in overweight or obese men and women aged 45-74 years with type 2 diabetes. The investigators propose to add validated and well-established measures of physical and cognitive performance to the year 8 follow-up visit - during the trial's weight maintenance phase - in ~1000 participants at 4 of the 16 Look AHEAD field sites (Colorado, Memphis, Pennington and Pittsburgh).

The specific aims of this ancillary study are: 1) To determine the long-term effects of a lifestyle intervention designed to achieve and maintain weight loss on physical function; and 2) To determine the long-term effects of a lifestyle intervention designed to achieve and maintain weight loss on cognitive function. In addition, the investigators hypothesize that in the intervention group, larger initial weight loss, better weight loss maintenance, and higher physical activity will be associated with better physical and cognitive function. The investigators also hypothesize that in the control group weight loss will be associated with worse physical and cognitive function than in those who are weight stable or who have gained weight.

The number of obese older adults is rising rapidly and there are few data to guide an evidence-based clinical response to their management. The results of this study will provide the first direct evidence of the role of long-term intentional weight loss on the maintenance of physical and cognitive function in older obese adults with diabetes. Since this study is being done as an ancillary study to an on-going trial it can be done in a timely and cost-efficient manner.

ELIGIBILITY:
Inclusion Criteria:

* The only inclusion criterion is that the participant is considered "active" at his/her Year 8 or Year 9 visit in the main study.

Exclusion Criteria:

* The only exclusion criterion is the person is not willing to participate in this ancillary study.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Kritchevsky, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Tennessee-Memphis, Memphis, Tennessee

REFERENCES:
- [Derived] Ip EH, Chen SH, Rejeski WJ, Bandeen-Roche K, Hayden KM, Hugenschmidt CE, Pierce J, Miller ME, Speiser JL, Kritchevsky SB, Houston DK, Newton RL, Rapp SR, Kitzman DW. Gradient and Acceleration of Decline in Physical and Cognitive Functions in Older Adults: A Disparity Analysis. J Gerontol A Biol Sci Med Sci. 2022 Aug 12;77(8):1603-1611. doi: 10.1093/gerona/glac109. PMID 35562076
- [Derived] Beavers KM, Leng I, Rapp SR, Miller ME, Houston DK, Marsh AP, Hire DG, Baker LD, Bray GA, Blackburn GL, Hergenroeder AL, Jakicic JM, Johnson KC, Korytkowski MT, Dorsten BV, Kritchevsky SB; Action for Health in Diabetes Movement and Memory Ancillary Study Research Group. Effects of Longitudinal Glucose Exposure on Cognitive and Physical Function: Results from the Action for Health in Diabetes Movement and Memory Study. J Am Geriatr Soc. 2017 Jan;65(1):137-145. doi: 10.1111/jgs.14478. Epub 2016 Sep 27. PMID 27676466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who enrolled in the main Look AHEAD study were eligible to participate in this ancillary study. Starting at year 8 clinic visits of the main study at 4 sites (Pennington, Denver, Pittsburgh, and Memphis) participants were asked if they would participate in this study (9/09-06/12). Those who agreed & consented were then enrolled.
Period: Overall Study
Arm/Group | Lifestyle Intervention | Diabetes Support and Education (DSE)
Started | 556 | 533
Completed | 551 | 530
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: 8 participants signed consent but did not return for ancillary visit
Groups:
- Intensive Lifestyle Intervention (ILI): Intensive Lifestyle Intervention that includes diet, physical activity, and behavior modification. The goal of the ILI intervention was for individuals to achieve and maintain a loss of at least 7% of initial body weight.
- Diabetes Support and Education (DSE): Diabetes Support and Education offers an educational program to participants focusing on diet, physical activity, and social support (information on behavioral strategies are not presented).
- Total: Total of all reporting groups
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE) | Total
Number analyzed (Participants) | 553 | 528 | 1081
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (6.8) | 59.1 (6.7) | 59.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 304 | 618
  Male | 239 | 224 | 463
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 110 | 108 | 218
  Non Hispanic White | 401 | 378 | 779
  Other/multiple | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Short Physical Performance Battery (SPPB) Score
Description: The Short Physical Performance Battery (SPPB) was administered to assess lower extremity physical performance and consisted of standing balance tasks (side-by-side, semi- and full-tandem stands for 10 seconds each), time to complete 5 repeated chair stands, and a 6-m walk to assess usual gait speed. Each of the three performance measures was assigned a score ranging from 0 (inability to perform the task) to 4 (the highest level of performance) and summed to create an SPPB score ranging from 0 to 12 (best). Assessed 8 or 9 years post-randomization in Look AHEAD parent Study.
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: Only participants who attended the ancillary clinic visit and were able to do the SPPB were included in the analysis (n=954)
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Intensive Lifestyle Intervention (ILI): Intensive Lifestyle Intervention includes diet, physical activity, and behavior modification. The goal of the ILI intervention was for individuals to achieve and maintain a loss of at least 7% of initial body weight.
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 486 | 468
Score on a scale | 10.1 (1.9) | 10.0 (2.1)

2. Secondary Outcome: Gait Speed Over 400 m
Description: A 400 m walk was administered to assess endurance. Participants were instructed to walk at their usual pace and time to complete the 400-m walk was recorded. The 400-m walk test was terminated if the participant reported chest pain, tightness or pressure, significant shortness of breath or difficulty breathing, feeling faint, lightheaded or dizzy, or other pain (e.g., leg pain).Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: Only participants who attended the ancillary clinic visit and were able to complete the 400 m walk were included in the analysis (n=869)
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 447 | 422
m/sec | 1.07 (.19) | 1.05 (.19)

3. Secondary Outcome: Grip Strength
Description: Grip strength (kg) was measured twice in each hand using an isometric Hydraulic Hand Dynamometer (Jamar, Bolingbrook, IL). The maximum of the force from two trials for the stronger hand was used in the analyses. Participants with severe hand pain or recent surgery in both hands were excluded from testing. Assessed 8 or 9 years post-randomization in Look AHEAD parent Study.
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: Only participants who attended the ancillary clinic visit and were able to do the grip strength test were included in the analysis (n=907)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 462 | 445
kg | 31 (10.2) | 30.7 (10.7)

4. Secondary Outcome: Knee Extensor Strength
Description: Maximum knee extensor strength (one repetition maximum (1RM)) was assessed on a Nautilus One™ Leg Extension machine. Participants with prior knee surgery on both knees where all or part of the joint was replaced were excluded from testing. The right leg was tested unless there was a contraindication (e.g., prior knee surgery). If participants experienced knee pain during the test and there were no contraindications to test the other leg, the other leg was tested; if participants experienced knee pain on the other leg, the test was terminated. Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: Only participants who attended the ancillary clinic visit and were able to achieve maximum knee extensor strength (1RM) were included in the analysis (n=701)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 359 | 342
kg | 23.4 (11.9) | 23.4 (12.5)

5. Secondary Outcome: Trail Making Test (Part A & B)
Description: Trail Making Tests A and B was used to assess attention and concentration (Part A) and executive function (Part B). Part A measures the time (in seconds) to draw lines to connect circled numbers in a numerical sequence and Part B measures the time (in seconds) to draw lines to connect circled numbers and letters in an alternating numeric and alphabetic sequence as rapidly as possible. The difference (in seconds; greater time indicates worse performance) in performance on Part B minus Part A was used in analysis to represent the contrast between performance on the simple (Part A) and alternating conditions (Part B). Assessed 8 or 9 years post-randomization in Look AHEAD parent Study.
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: Only participants who attended the ancillary clinic visit and completed the cognitive battery were included in the analysis (n=978)
Measure: Mean (Standard Deviation); unit: secs
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 499 | 479
secs | 62.87 (46.14) | 62.85 (46.34)

6. Secondary Outcome: Digit Symbol Substitution Test (DSST)
Description: The Digit Symbol Substitution Test (DSST) was used to assess working memory. Participants were presented with a legend at the top of the page showing the boxes each with a number from 1 to 9 and below each numbered box is a unique symbol. As rapidly as possible, the participant fills in the randomly ordered boxes with numbers paired with blank boxes with the symbol that corresponds to the number in the legend. The score is the total number of correctly entered symbols completed in 90 seconds (range, 0-133; higher score indicates better performance). Assessed 8 or 9 years post-randomization in Look AHEAD parent Study.
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 499 | 479
number correct | 41.61 (10.38) | 41.14 (10.84)

7. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: The Rey Auditory Verbal Learning Test (RAVLT) was used to assess verbal memory. The participant is read a list of 15 words five times. After each time the list is given, the participant is asked to immediately recall as many words as possible. Following the fifth recall, an interference list is presented, after which the participant is asked to spontaneously recall words from the original list. After a 10-minute interval has passed, the participant is asked again to recall as many words as possible from the original list. The number of words correctly recalled on the delayed recall were used in the analysis (range, 0-15; higher number correct indicates better performance). Assessed 8 or 9 years post-randomization in Look AHEAD parent Study.
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 499 | 479
number correct | 7.51 (3.28) | 7.30 (3.22)

8. Secondary Outcome: Modified Stroop Color and Word Test
Description: The Modified Stroop Color and Word Test was used to assess executive function. The test measures a participant's ability to view complex visual stimuli and to respond to one stimulus dimension while suppressing response to another competitive stimulation. The participant first reads aloud words denoting colors printed in black ink (Subtest 1), then names aloud the color of blocks printed in colored ink (Subtest 2), and finally names aloud the color ink in which the words are printed in which are incongruent to the word (Subtest 3). The amount of time to complete each subtest and the number of errors are recorded and interference calculated as time to complete Subtest 3 - Subtest 1 + errors (lower interference scores indicate better cognitive performance). Assessed 8 or 9 years post-randomization in Look AHEAD parent Study.
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 499 | 479
score on a scale | 39.17 (17.71) | 38.47 (18.68)

9. Secondary Outcome: Modified Mini-Mental Status Exam (3MS)
Description: The Modified Mini-Mental Status Exam (3MS) was used to assess global cognitive function. Scores range from 0 to 100 with higher scores indicating better cognitive function. Assessed 8 or 9 years post-randomization in Look AHEAD parent Study.
Time Frame: Assessed 8 or 9 years post-randomization in Look AHEAD parent Study
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intensive Lifestyle Intervention (ILI) | Diabetes Support and Education (DSE)
Number analyzed (Participants) | 499 | 479
Score on a scale | 92.25 (5.94) | 92.19 (6.66)

ADVERSE EVENTS:
Time Frame: 1-2 weeks
Arm/Group | Lifestyle Intervention | Diabetes Support and Education (DSE)
Serious Adverse Events (participants affected / at risk) | 0/556 | 0/533
Other Adverse Events (participants affected / at risk) | 0/556 | 0/533

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No